CLINICAL TRIAL: NCT07369713
Title: Efficacy and Safety of Accelerated Intermittent Theta-burst Stimulation (a-iTBS) in Adolescents With Depression: A Randomized, Double-Blind, Controlled Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1stChongqingCQMU___ZXYa-iTBS
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment design. Participants will be randomly assigned in a 1:1:1 ratio to the experimental target a-iTBS treatment group, the conventional target a-iTBS treatment group, or the sham stimulation group. All three groups will utilize the Blackdolphin TMS Robot device (SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., receiving 50 sessions of a-iTBS stimulation (5 Hz, 90% RMT) or sham stimulation over 10 consecutive days, with consistent intervention frequency and procedures. Participants will remain in their assigned group for the entire study duration without any crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental target a-iTBS treatment group (Experimental): Participants will undergo MRI-guided identification of the voxel in the left dorsolateral prefrontal cortex (DLPFC) that is most negatively correlated with the functional connectivity of the subgenual anterior cingulate cortex (sgACC) as the stimulation site. Accelerated Intermittent Theta-burst Stimulation (a-iTBS) (5 Hz, 90% RMT) will be administered using the Blackdolphin TMS Robot device (model SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., with 50 sessions over 10 consecutive days.
  Interventions: Device: Experimental target a-iTBS treatment
- Conventional target a-iTBS treatment group (Experimental): Participants will undergo MRI-guided identification of the standard F3 target in the dorsolateral prefrontal cortex (DLPFC) as the stimulation site. Accelerated Intermittent Theta-burst Stimulation (a-iTBS) (5 Hz, 90% RMT) will be administered using the Blackdolphin TMS Robot device (model SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., with 50 sessions over 10 consecutive days.
  Interventions: Device: Conventional target a-iTBS treatment
- Sham stimulation treatment group (Sham Comparator): Participants will receive a sham stimulation treatment designed to simulate the a-iTBS procedure without generating an effective magnetic field output. The intervention will use a dedicated sham stimulation coil, which is identical in appearance, operation, and stimulation protocol to the experimental group. This coil is designed to maintain the same auditory and tactile sensations as the active stimulation but is equipped with an electromagnetic shielding structure or an internal reverse coil arrangement to effectively prevent magnetic flux from penetrating the skull, ensuring no actual neuromodulatory effects.
  Interventions: Device: Sham stimulation treatment

INTERVENTIONS:
Device: Experimental target a-iTBS treatment — Participants will undergo MRI-guided identification of the voxel in the left dorsolateral prefrontal cortex (DLPFC) that is most negatively correlated with the functional connectivity of the subgenual anterior cingulate cortex (sgACC) as the stimulation site.
  Arms: Experimental target a-iTBS treatment group
Device: Conventional target a-iTBS treatment — Participants will undergo MRI-guided identification of the standard F3 target in the dorsolateral prefrontal cortex (DLPFC) as the stimulation site.
  Arms: Conventional target a-iTBS treatment group
Device: Sham stimulation treatment — Participants will receive a sham stimulation treatment designed to simulate the a-iTBS procedure without generating an effective magnetic field output.
  Arms: Sham stimulation treatment group

SUMMARY:
This study aims to assess the feasibility, safety, acceptability, and preliminary efficacy trends of a Accelerated Intermittent Theta-burst Stimulation (a-iTBS) intervention for adolescent depression through a pilot clinical trial. The findings will inform the design and optimization of subsequent formal randomized controlled trials, providing essential evidence for their execution.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled pilot trial aimed at evaluating the feasibility, safety, acceptability, and preliminary efficacy trends of Accelerated Intermittent Theta-burst Stimulation (a-iTBS) for the treatment of adolescent depression.

Adolescents diagnosed with Major Depressive Disorder (MDD) will be randomly assigned in a 1:1:1 ratio to one of three groups: the experimental target a-iTBS treatment group, the conventional target a-iTBS treatment group, and the sham stimulation group. All three groups will receive 10 consecutive days of a-iTBS stimulation (5 Hz, 90% RMT) or sham stimulation intervention, using the Blackdolphin TMS Robot (SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., with 50 sessions in total. The intervention frequency and procedure will remain consistent across all groups.

In the experimental target a-iTBS treatment group, participants will undergo MRI-guided identification of the left dorsolateral prefrontal cortex (DLPFC) region, where the voxel most negatively correlated with the functional connectivity of the subgenual anterior cingulate cortex (sgACC) will serve as the stimulation target. In the conventional target a-iTBS treatment group, participants will have the standard F3 target in the DLPFC identified via MRI guidance as the stimulation site. Participants in the sham stimulation group will receive a placebo treatment, simulating the a-iTBS procedure without generating an effective magnetic field output.

The primary outcome of the treatment phase is the efficacy rate or the remission rate of depressive symptoms. Secondary outcomes include symptom scales, anxiety symptoms, suicide risk, quality of life, sleep, rumination, and cognition. Safety will be monitored through adverse events, vital signs, laboratory tests, and tolerability assessments.

ELIGIBILITY:
Inclusion Criteria:

(1) Age 12 - 18 (2) Diagnosis of major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), confirmed through the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime version (K-SADS-PL), currently in a depressive episode (3) Score≥40 on the CDRS-R (4) Stable pharmacological treatment: At least 4 weeks of stable psychiatric medication use prior to enrollment, with continuation of the same psychiatric medication regimen throughout the study.

-

Exclusion Criteria:

1. Psychiatric comorbidities other than anxiety disorders
2. Depression with psychotic symptoms
3. Young Mania Rating Scale (YMRS) score >13
4. A history of neurological disorders (e.g., epilepsy, brain injury) or severe somatic diseases (e.g., thyroid disorders, lupus, diabetes, pulmonary, hepatic, or renal impairment, major trauma)
5. Patients currently using anticonvulsants or high-dose benzodiazepines
6. A history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or other neuromodulation treatments
7. A history of alcohol or substance abuse or dependence
8. Women who are pregnant or breastfeeding
9. Current high suicide risk
10. Potential complicating factors related to transcranial magnetic stimulation, such as scalp conditions or perforations that may affect magnetic field delivery
11. Contraindications to MRI -

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in CDRS-R (Children's Depression Rating Scale) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Response rate of depressive symptoms (defined as ≥50% reduction in CDRS-R score) or remission rate of depressive symptoms (defined as CDRS-R score ≤28).

SECONDARY OUTCOMES:
Change in BDI-II (Baker Depression Scale) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Change in BDI-II (Baker Depression Scale) scores from baseline
Change in SCARED (The Screen for Child Anxiety-Related Emotional Disorders) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Improvement in anxiety (SCARED minus the scores）
Change in suicide risk from baseline on the C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  The severity of the suicide risk
Change in PSQI (Pittsburgh Sleep Quality Index) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Improvement in sleep status (PSQI minus the scores）
Change in PedsQL4.0 (The Pediatric Quality of Life Inventory) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Improvement of children's quality of life（PedsQL4.0 minus the scores)
Change in CGI-S (Clinical Global Impressions-Severity Scales) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Improvement in overall clinical impression severity（7-point scale, with 1 being normal and 7 being among the most severely damaged）
Change in CGI-I (Clinical Global Impressions-Improvement Scales) scores from baseline | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  Improvement of clinical general Impression scale（ 7-point scale,7 denoting a very significant deterioration）
Change in RSS (Ruminative Responses Scale) | Baseline of treatment period, 10 days; The follow-up period was 1 month, 3 months
  The level of improvement in negative thinking（The higher the total score, the more reflective thinking The more severe it is）

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China